CLINICAL TRIAL: NCT05234047
Title: Observational Study Evaluating the Effect of a Biotherapy Treatment (Anti- RANKL Ligand Antibody: Denosumab) on Bone and Vascular Metabolism in Osteoporotic Chronic Kidney Disease Patients
Brief Title: Study Evaluating Denosumab on Vascular and Bone Metabolism in Osteoporotic Chronic Kidney Disease (HDENOBS)
Acronym: HDENOBS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL21_0451
Record Dates: First submitted 2022-01-31; First posted 2022-02-10 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Osteoporosis; Chronic Kidney Disease 5D
MeSH Terms: conditions — Osteoporosis | interventions — Absorptiometry, Photon

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CKD-5D patients receiving denosumab
  Interventions: Procedure: MDCT (multidetector computed tomography); Procedure: Dual-energy X-ray absorptiometry

INTERVENTIONS:
Procedure: MDCT (multidetector computed tomography) — MDCT will be performed at inclusion and after 2 years
Procedure: Dual-energy X-ray absorptiometry — DXA will be performed at inclusion, 1 and 2 years after inclusion

SUMMARY:
Aim of this study is to evaluate in a population of osteoporotic chronic kidney disease patients the effect of denosumab:

* on coronary artery calcification scores evolution after 24 months of followup
* on abdominal aorta calcification scores evolution after 24 months of followup
* on bone mineral density (femoral T-score) at 24 months
* on bone mineral density evolution (femoral T-score) after 24 months of follow-up
* on bone mineral density evolution (lumbar T-score) after 24 months of follow-up
* on parameters of bone remodelling after 24 months of follow-up
* on cardiovascular morbidity (cardiovascular events) and mortality after 24 months of follow-up
* the tolerance after 24 months of follow-up

DETAILED DESCRIPTION:
Aim of this study is to evaluate in a population of osteoporotic chronic kidney disease patients the effect of denosumab:

* on coronary calcification scores evolution (by multidetector computed tomography) after 24 months of follow-up
* on abdominal aorta calcification scores evolution (by plain abdominal Xray) after 24 months of follow-up
* on bone mineral density (femoral T-score) (by bone densitometry) at 24 months
* on bone mineral density evolution (femoral T-score) (by bone densitometry) after 24 months of follow-up
* on bone mineral density evolution (lumbar T-score) (by bone densitometry) after 24 months of follow-up
* on parameters of bone remodelling after 24 months of follow-up
* on cardiovascular morbidity (cardiovascular events) and mortality after 24 months of follow-up
* the tolerance after 24 months of follow-up

ELIGIBILITY:
Inclusion Criteria:

* Chronic kidney disease stage 5D patient, hemodialyzed with extracorporeal treatment for at least 3 months
* Osteoporosis

Exclusion Criteria:

* Pregnancy or breastfeeeding female
* Current corticoid treatment
* PTH and Calcium outside the KDIGO guidelines
* Adynamic bone disease suspicion
* Cancer or myeloma
* Serious hepatic cytolysis
* Serious dental troubles
* Positive HIV serology
* Hypersensibility to active substance or one of excipients of denosumab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: CKD-5D patients with osteoporosis
Sampling Method: Non-Probability Sample
Enrollment: 21 (Estimated)
Dates: Start 2022-05 (Estimated); Primary Completion 2025-02 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Relative variation of coronary calcification scores after 24 months of follow-up | 24 months after inclusion

SECONDARY OUTCOMES:
Relative variation of abdominal aorta calcification scores after 24 months of follow-up | 24 months after inclusion
Relative variation of femoral bone mineral density after 24 months of follow-up (T-score evaluated by osteodensitometry) | 24 months after inclusion
Relative variation of lumbar bone mineral density after 24 months of follow-up (T-score evaluated by osteodensitometry) | 24 months after inclusion
Relative variation of radius bone mineral density after 24 months of follow-up (T-score evaluated by osteodensitometry) | 24 months after inclusion
Relative variation of whole body bone mineral density after 24 months of follow-up (T-score evaluated by osteodensitometry) | 24 months after inclusion
Variation of calcium at 6, 12, 18 and 24 months of follow-up | 6, 12, 18 and 24 months after inclusion]
Variation of phosphorus at 6, 12, 18 et 24 months of follow-up | 6, 12, 18 and 24 months after inclusion
Variation of bone remodeling at 6, 12, 18 et 24 months of follow-up | 6, 12, 18 and 24 months after inclusion
Variation of inflammation at 6, 12, 18 et 24 months of follow-up | 6, 12, 18 and 24 months after inclusion
Morbi-mortality at 24 months of follow-up | 24 months after inclusion]
Adverse events occuring during the entire study | 24 months after inclusion]